CLINICAL TRIAL: NCT02663726
Title: A Pilot Randomised Controlled Trial Investigating the Effects of a 10-week Yoga Intervention on Physical Function and Health-related Quality of Life in Physically-inactive Older Adults
Brief Title: Adapted Yoga for Inactive Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Yorkshire Yoga & Therapy Centre (Unknown); The British Wheel of Yoga (Unknown); Big Lottery Fund - Awards for All (Unknown)
Responsible Party: Principal Investigator, Garry Tew, Reader in Exercise and Health Sciences, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLSGT180116
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: The Study Will Recruit Adults Aged 60 Years or Older
Keywords: Physically inactive; Older adults
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga intervention group (Experimental): 10 weekly 75-min sessions of specialised yoga plus written advice about physical activity for older adults
  Interventions: Other: Yoga; Behavioral: Written advice
- Waiting list control group (Active Comparator): Usual care plus written advice about physical activity for older adults
  Interventions: Behavioral: Written advice

INTERVENTIONS:
Other: Yoga — 10 weekly 75-min sessions of specialised yoga
  Arms: Yoga intervention group
Behavioral: Written advice — Written advice about physical activity

SUMMARY:
There is evidence that yoga has beneficial effects on several aspects of physical and mental health. However, few studies have explored the acceptability and health effects of yoga in older adults. This preliminary study will explore the effects of a 10-week yoga intervention on physical function and quality of life in older adults. Data collected in this study will be used to inform the design of a subsequent adequately-powered randomised controlled trial.

DETAILED DESCRIPTION:
Older adults (i.e. aged ≥60 years) who are physically inactive are at increased risk of falls, functional limitations, disability, and mental health problems. Encouragingly, there is evidence that various physical activity interventions can elicit meaningful improvements in physical function and health-related quality of life in older people. Effective programmes have included aerobic exercise, progressive resistance training and Tai Chi. Yoga is an alternative approach to improving fitness and health outcomes in older adults. The benefits of yoga may be greater than those of exercise alone because yoga offers a combination of physical exercise with mental focus, and participants are taught good posture, self-awareness, and self-care along with relaxation. Indeed, a recent systematic review and meta-analysis that included 16 studies (n=649) concluded that yoga may provide greater improvements in physical functioning and self-reported health status than conventional physical activity interventions in elderly people. However, the previous studies had limitations, including small sample sizes, a single yoga teacher delivering the programme, and short-term follow-up. Furthermore, none of the included studies had been conducted in the United Kingdom. Many different schools of hatha yoga exist in the West, such as Iyengar, Sivananda, Viniyoga, Bikram (Hot Yoga), and it is likely that some of these forms are more acceptable and effective than others in elderly people, many of whom present with multiple morbidities. Gentle Years Yoga© is a yoga programme which was developed in North Yorkshire, England by the British Wheel of Yoga 'Approved Centre' Yorkshire Yoga in 2009 to cater specifically for the needs of older people with age-related conditions such as osteoarthritis, arthroplasty, dementia, sensory impairment. To date, only anecdotal evidence exists regarding the acceptability, feasibility and effectiveness of this programme; therefore, further research is warranted. Here, we are proposing to conduct a two-arm, parallel-group, pilot randomised controlled trial in physically inactive adults aged ≥60 years, the aims of which are to: (i) inform the design of, and assess the feasibility of conducting, a definitive randomised controlled trial, and; (ii) explore the acceptability, safety and potential benefits of the Gentle Years Yoga© programme in this specific population.

ELIGIBILITY:
Inclusion Criteria:

Age ≥60 years Able to provide written informed consent and complete the study questionnaires Able to travel to a study centre for assessment visits and yoga sessions

Exclusion Criteria:

Absolute contraindications to exercise testing and training as defined by the American College of Sports Medicine Planned major surgery within 3 months of the proposed baseline assessment date Current participation in >90 min/week of purposeful exercise, such as jogging or swimming Participation in another clinical trial for with concurrent participation is deemed inappropriate

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Short Performance Physical Battery | 3 months

SECONDARY OUTCOMES:
EQ-5D-5L | 3 months
Warwick-Edinburgh Mental Well-being Scale | 3 months
Back scratch test of upper-body flexibility | 3 months
Chair sit-and-reach test of lower-body flexibility | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Garry A Tew, PhD, Principal Investigator — Northumbria University
Locations (1):
- Yorkshire Yoga & Therapy Centre, Knaresborough, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel NK, Newstead AH, Ferrer RL. The effects of yoga on physical functioning and health related quality of life in older adults: a systematic review and meta-analysis. J Altern Complement Med. 2012 Oct;18(10):902-17. doi: 10.1089/acm.2011.0473. Epub 2012 Aug 21. PMID 22909385
- [Background] Youkhana S, Dean CM, Wolff M, Sherrington C, Tiedemann A. Yoga-based exercise improves balance and mobility in people aged 60 and over: a systematic review and meta-analysis. Age Ageing. 2016 Jan;45(1):21-9. doi: 10.1093/ageing/afv175. Epub 2015 Dec 25. PMID 26707903
- [Derived] Tew GA, Howsam J, Hardy M, Bissell L. Adapted yoga to improve physical function and health-related quality of life in physically-inactive older adults: a randomised controlled pilot trial. BMC Geriatr. 2017 Jun 23;17(1):131. doi: 10.1186/s12877-017-0520-6. PMID 28645259